CLINICAL TRIAL: NCT03143985
Title: A Phase 1b Trial of Vactosertib in Combination With Pomalidomide (POM) in Relapsed or Relapsed and Refractory Multiple Myeloma (RRMM)
Brief Title: Vactosertib in Combination w/ Pomalidomide in Relapsed or Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Koen van Besien (Other)
Responsible Party: Sponsor-Investigator, Koen van Besien, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A17
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Vactosertib; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — vactosertib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vactosertib + Pomalidomide (Experimental): Vactosertib tablets, taken once daily for the first and second dose levels and twice a day for third and fourth dose level levels for 5 days followed by 2 days without treatment, repeated for 28-day cycles until evidence of progressive disease, intolerable toxicity, or participant discontinuation.
  For dose escalation - dosing initiated at 60 mg once daily by oral administration and will be increased to determine MTD. Provisional subsequent doses are 60, 120, once daily and 100 mg and 200 mg twice daily on days 1-5, 8-12, 15-19 and 22-26. Extension cohorts will enter at 200 mg twice daily (i.e. if MTD not defined) for 12 months until progression or intolerable toxicity.
  POM is administered orally (4 mg/day daily on Days 1 - 21 days). Treatment will occur in a suitable outpatient ambulatory care setting that is equipped for monitoring of patients with hematopoietic malignancies undergoing early clinical trial research.
  Interventions: Drug: Vactosertib; Drug: Pomalidomide

INTERVENTIONS:
Drug: Vactosertib — Vactosertib is an inhibitor of protein serine/threonine kinase activity of TGF-β receptor type 1 (TGFBR1; ALK5). Vactosertib inhibits the phosphorylation of the ALK5 substrates, Smad2 and Smad3, and the intracellular signaling of TGF-β. Dosing begins at 60mg by mouth, daily and may increase to 240mg by mouth daily in the absence of dose limiting toxicities
  Other Names: TEW-7197; EW7197; EW-7197
Drug: Pomalidomide — POM, an analog of thalidomide, is an immunomodulatory agent with antineoplastic activity. Myeloma tumor cells exposed to POM, undergo growth arrest and increased apoptotic cell death. POM enhances T cell- and natural killer cell-mediated immunity and inhibit production of pro-inflammatory cytokines by monocytes. POM may be taken orally with water. Capsules should not be broken, chewed or opened. POM should be taken without food (at least 2 hours before or 2 hours after a meal). POM will be commercially available. POM will be taken by mouth at a dose of 4mg per day
  Other Names: POM

SUMMARY:
The purpose of this study is to see if the study drug, called Vactosertib, is safe and determine what the best dose is to treat future patients when given in combination with pomalidomide (POM). The study will also look to see if it has any effect on multiple myeloma, when given in combination with POM.

DETAILED DESCRIPTION:
Primary Objective

* To determine the maximum tolerated dose (MTD) or maximum tested dose level of Vactosertib given in combination with pomalidomide (POM) for the treatment of relapsed or relapsed or refractory multiple myeloma (RRMM)
* To characterize the safety and tolerability profile of Vactosertib in combination with POM at the MTD

Secondary Objectives

To evaluate the activity of the combination of Vactosertib/POM regimen in terms of:

* Overall response rate (complete response [CR] + very good partial response [VGPR] +partial response [PR]) and clinical benefit rate (CR + VGPR + PR + minimal response [MR]) based on International Myeloma Working Group (IMWG) defined response criteria and the duration of response (DOR) in RRMM patients.
* Progression-free survival (PFS) and PFS at 6 months (PFS-6)

Exploratory Objective:

To evaluate the bone remodeling and immunologic effects of POM/Vactosertib combination therapy and its correlation with clinical outcome in patients with multiple myeloma.

Study Design To evaluate the bone remodeling and immunologic effects of POM/Vactosertib combination therapy and its correlation with clinical outcome in patients with multiple myeloma. This study is a Phase I, open label trial of Vactosertib in combination with standard doses of POM. The study will be conducted as a modified Fibonacci 3 + 3 dose escalation design to determine the MTD of Vactosertib in combination with standard doses of POM. Patients will receive combination Vactosertib/POM.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given voluntary written informed consent before performance of any study-related procedures not part of standard (non-investigational) medical care.
* Patient has been previously diagnosed with multiple myeloma based on standard criteria.
* Patient has relapsed or refractory disease according to international uniform response criteria and must have previously received therapy with:

  * A proteasome inhibitor and Immunomodulatory imide drugs (IMiD)
  * All subjects must have documented disease progression during or after their last antimyeloma therapy.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2.
* Patient has measurable disease defined as at least one of the following:

  * Serum M protein ≥ 0.5 /dL (≥5 g/L)
  * Urine M protein ≥ 200 mg/24 hours
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
* Clinical Laboratory Inclusion Criteria: The following laboratory results must be met within 14 days (or as stipulated) prior to study drug (treatment) administration:

  * Absolute neutrophil count (ANC) ≥ 1000 cells/μl (growth factor cannot be used within the previous 5 days)
  * Platelet count ≥ 50,000/μl (without platelet transfusion in the previous 5 days)
  * Aspartate aminotransferase (AST/SGOT) and Alanine aminotransferase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN)
  * Serum total bilirubin ≤ 2.0 mg/dL or >3.0 x ULN for subjects with hereditary benign hyperbilirubinemia
  * Creatinine clearance ≥ 30 ml/min (calculated by the Cockcroft-Gault Equation or per 24 hour urine collection)
  * Serum calcium (corrected for albumin) level at or below the ULN range (treatment of hypercalcemia is allowed and subject may enroll if hypercalcemia returns to normal range with standard treatment).
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test prior to initiation of the study treatment with Vactosertib/POM. The test must have a sensitivity of at least 50 mIU/mL. Study participants who are FCBP must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking POM through 30 days after the last dose of POM and 60 days after the last dose of Vactosertib. FCBP must also agree to ongoing pregnancy testing during the entire duration of treatment. Men must agree to use a latex or synthetic condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 60 days after the last dose of POM or Vactosertib. These same patients must not donate sperm. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. All patients enrolled into this trial, must agree to be registered in and must comply with all requirements of the Pomalidomide Risk Evaluation and Mitigation Strategy (POM REMS™) program.

Exclusion Criteria:

* Prior therapy with Vactosertib or received any investigational drug within the prior 28 days.
* Plasma Cell Leukemia
* Patients with solitary plasmacytoma
* Patients who are primarily eligible for autologous stem cell transplant
* Prior anti-cancer therapy (chemotherapy, targeted agents, radiotherapy, and immunotherapy) within the prior 21 days except for alkylating agents (e.g., melphalan) within the prior 28 days.
* Prior treatment with pomalidomide.
* Subjects with active malignancy and/or cancer history that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the trial collaborator, MedPacto Inc., before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including superficial bladder cancer), cervical intraepithelial neoplasia, and organ-confined prostate cancer with no evidence of progressive disease
* Any > grade 1 (according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE) v.4.03) adverse reaction unresolved from previous treatments or not readily managed and controlled with supportive care. The presence of alopecia of any grade and peripheral neuropathy ≤ Grade 2 without pain is allowed.
* Previous allogeneic stem cell transplantation with active graft versus host disease (GVHD), or treatment with immunosuppressive therapy in the 2 months prior to study entry.
* No oral corticosteroids 3 days before initiating combinations Vactosertib/POM; inhaled corticosteroids are permitted.
* Patient is known to be human immunodeficiency virus (HIV) positive, or have chronic or active Hepatitis B (core- or surface antigen-positive) or active hepatitis C infection.
* Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association (NYHA) Class 3 or 4, congestive heart failure, uncontrolled or unstable angina, history of myocardial infarction or stroke within 6 months prior to study entry, or clinically significant arrhythmias not controlled by medication).
* Major abnormalities identified by ECG or echocardiogram (ECHO), at the Investigator's discretion.
* Presence of aneurisms of the ascending aorta or aortic stress.
* Hypertension that is not controlled by standard medication (to 150/90 mmHg or below).
* Uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), pulmonary hypertension) that in the opinion of the investigator would put the patient at significant risk for pulmonary complications during the study.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation (DIC), or psychiatric illness/social situations that would limit compliance with study requirements.
* History of erythema multiforme or severe hypersensitivity to prior IMiD's such as thalidomide and lenalidomide.
* Patients requiring hemodialysis
* The patient is receiving medications that are:

  * Exclusively or primarily eliminated by cytochrome P-450 isozyme 3A4 (CYP3A4).
  * Exclusively or primarily eliminated by Uridine 5'-diphospho (UDP)-glucuronyltransferase 1A1 (UGT1A1).
  * Substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window; or which are strong inhibitors of drug transporter MDR1.
* Patients should have discontinued strong CYP1A2 inhibitors (e.g. ciprofloxacin and fluvoxamine) at least five half-lives before beginning study treatment.
* Inability to tolerate thromboprophylaxis (Required Concurrent Medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or maximum tested dose level of Vactosertib given in combination with POM for the treatment of relapsed or RRMM | Up to 30 days after treatment ends (24 weeks + 30 days)
  the largest tested dose where multiple dose limiting toxicities are not observed

SECONDARY OUTCOMES:
Overall response rate | Up to 6 months after beginning treatment
  overall response is the complete response [CR] + very good partial response [VGPR] + partial response [PR] based on International Myeloma Working Group (IMWG) defined response criteria
Progression-free survival (PFS) | Up to 30 days after discontinuation of treatment
  Progression-free survival will be measured from study entry to progression or death of any cause, whichever comes first.
Progression-free survival at 6 months (PFS-6) | Up to 6 months after beginning treatment
  Number of patients who did not progress on treatment, at 6 months after beginning treatment
Duration of Response | Up to 6 months after beginning treatment
  The time from the first confirmed response to progression of disease. Responses include Complete Response (CR), Stringent CR, Very Good Partial Response, Partial Response, Minor Response, Stable disease. Responses based on International Myeloma Working Group (IMWG) defined response criteria
clinical benefit rate | Up to 6 months after beginning treatment
  clinical benefit rate is the CR + VGPR + PR + minimal response [MR] based on International Myeloma Working Group (IMWG) defined response criteria
Overall Survival | Up to 6 months after progression
  Overall survival for all will be measured from study entry to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Koen van Besien, MD, PhD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Malek E, Rana PS, Swamydas M, Daunov M, Miyagi M, Murphy E, Ignatz-Hoover JJ, Metheny L, Kim SJ, Driscoll JJ. The TGFbeta type I receptor kinase inhibitor vactosertib in combination with pomalidomide in relapsed/refractory multiple myeloma: a phase 1b trial. Nat Commun. 2024 Aug 27;15(1):7388. doi: 10.1038/s41467-024-51442-2. PMID 39191755